CLINICAL TRIAL: NCT04489810
Title: GlutDigest - Enzymes-assisted Gluten Digestion
Brief Title: Digestion of Gluten in the Presence of Enzymes
Acronym: GlutDigest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Archer-Daniels-Midland Company (Industry)
Collaborators: Teagasc (Industry); Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Project 0470
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-05

CONDITIONS: Main Focus: Gluten and Starch Digestibility
Keywords: Gluten; Starch; Digestive enzymes; Probiotics

STUDY DESIGN:
Intervention Model Description: Each participant attended a clinic for one day for an acute assessment of the acute effects of treatment. This was done on the same day over 4 consecutive weeks. At each visit the participant received 1 of 4 different treatments
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Meal A + Placebo (Placebo Comparator): 350 mg Placebo capsule, taken by mouth, once, with Meal A
  Interventions: Dietary Supplement: Placebo; Other: Meal A
- Meal A + Elevase® (Experimental): 350 mg Elevase® capsule, taken by mouth, once, with Meal A
  Interventions: Dietary Supplement: Elevase®; Other: Meal A
- Meal A + DE111® (Experimental): 350 mg DE111® capsule, taken by mouth, once, with Meal A
  Interventions: Dietary Supplement: DE111®; Other: Meal A
- Meal B + Placebo (Experimental): 350 mg Placebo capsule, taken by mouth, once, with Meal B
  Interventions: Dietary Supplement: Placebo; Other: Meal B

INTERVENTIONS:
Dietary Supplement: Placebo — Maltodextrin capsule manufactured to mimic the Elevase® and DE111® capsules
  Arms: Meal A + Placebo; Meal B + Placebo
Dietary Supplement: Elevase® — 1 capsule containing 350 mg of Elevase®
  Arms: Meal A + Elevase®
Dietary Supplement: DE111® — 1 capsule containing Bacillus subtilis DE111
  Arms: Meal A + DE111®
Other: Meal A — Oatmeal porridge - serving of cooked oats containing 50g of carbohydrates (excluding sugars); Wheat cereal - serving of wheat cereal providing 1g of gluten; Water - 125 mL
  Arms: Meal A + DE111®; Meal A + Elevase®; Meal A + Placebo
Other: Meal B — Refrigerated oatmeal - serving of refrigerated oats containing 50g of carbohydrates (excluding sugars); Wheat cereal - serving of wheat cereal providing 1g of gluten; Water - 125 mL
  Arms: Meal B + Placebo

SUMMARY:
This study evaluates the impact of two dietary supplements (Elevase® and DE111®) and of oatmeal properties on the digestion of gluten and starch and on the glycemic response.

DETAILED DESCRIPTION:
RATIONALE Two important factors can influence the proportions of gluten and starch that resist digestion: (1) enzyme availability and specificity and (2) the structural properties of the food.

Elevase®, is a dietary supplement based on an enzyme preparation which effectively degrades gluten in vitro (Healey, Hall et al. unpublished). As it has also been found that the rate of wheat protein digestion can be increased in the presence of amylases (Smith, Pan et al. 2015), Elevase® is also enriched with amylase to aid in starch digestion.

The structural properties of food are influenced by numerous factors including meal preparation practices. Two common practices that can influence nutrient availability differently are heating vs. refrigerating (e.g. oat porridge vs. soaked and refrigerated oats).

Bacillus subtilis DE111® can produce and secrete many enzymes, including proteases, which, if secreted into the environment of the digestive tract, could support digestion and, in particular, the digestion of gluten. However, it is not clear whether diet supplementation with DE111 is a physiologically viable approach in terms of probiotic survival in the gastrointestinal tract.

PURPOSE The aims of this study are to better understand the impact of each of these factors and whether supplementation with probiotic spores is a viable option.

ELIGIBILITY:
Inclusion Criteria:

* Subject has given written informed consent
* Subject has an ileostomy stable for at least 3 months post-operative and shows normal stoma functions
* Subject is otherwise healthy
* Subject is available to participate in the study sessions on the proposed dates

Exclusion Criteria:

* Subject has coeliac disease or allergy to wheat products and/or any other ingredients in the test meal and standard meals
* Case of obstruction of the stoma in the past 3 months
* Body mass index < 18 kg/m2 or > 30 kg/m2.
* Diagnosed mouth, throat or active gastrointestinal pathology (other than ileostomy) that may affect normal ingestion and digestion of food.
* History of pancreatic disease
* Subject is immunocompromised (HIV positive, transplant patient, on antirejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy within the last year)
* Subject has Type 1 or Type 2 diabetes mellitus.
* Subject has a history of bariatric surgery.
* Subject has a history of drug and/or alcohol abuse at the time of enrolment
* Subject is currently participating in another study, or plans to participate in another study during the study period
* Women of child-bearing potential who do not use an acceptable method of contraception
* Pregnant or nursing (lactating) women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Undigested wheat protein | 9-hour period after the test meal
  Difference between the mean concentration of undigested wheat protein in ileal effluent samples.

SECONDARY OUTCOMES:
Vegetative DE111 cells | 9-hour period after the test meal
  Mean concentration of DE111® cells recovered in the ileal effluent in the vegetative state.
Glycemic response | At baseline, and at different time-points during 9 hours after after consuming the test meal.
  Difference between the mean area under the glucose concentration (measured in the interstitial fluid) curves following each treatment
Undigested starch | At baseline and once every hour in the 9-hour period after consumption of the test meal.
  Difference between the mean concentration of undigested starch in ileal effluent samples.
Undigested food particles | 9-hour period after the test meal
  Pictures of undigested foods particles and microscopy will be combined for a combined assessment of macro- and micro- structural characteristics of the food particles recovered in ileal effluent samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Food Clinical Trials, Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith F, Pan X, Bellido V, Toole GA, Gates FK, Wickham MS, Shewry PR, Bakalis S, Padfield P, Mills EN. Digestibility of gluten proteins is reduced by baking and enhanced by starch digestion. Mol Nutr Food Res. 2015 Oct;59(10):2034-43. doi: 10.1002/mnfr.201500262. Epub 2015 Aug 21. PMID 26202208